CLINICAL TRIAL: NCT04380194
Title: Detection of Intracorporeal Bioresistant Nanocomposites Tracing Short- and Long-term Neurological Disorders in a Collective Fulguration
Brief Title: Intracorporeal Nanocomposites and Neurological Disorders in Fulgurates (FulgurnanoF)
Acronym: Fulgurnano
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: PROMES UPR 8521 DR2-CNRS (Unknown); LPC UMR 6533, Campus Universitaire des Cézeaux (Unknown)
Responsible Party: Sponsor
Other Study IDs: RBHP 2018 CAUMONT; 2018-A01725-50 (Other: ANSM)
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Neurologic Disorder
Keywords: neurologic disorders; Keraunopathology; neuropsychological disorders; bioresistant nanocomposite; collective lightning-strike injuries
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Recovery of the bottoms of the victims' blood and urine tubes at H+4. Blood and urine samples from the victims at two years of age. Single blood and urine samples from the witnesses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- victims: thirteen patients affected by lightning in collective fulguration
  Interventions: Diagnostic Test: nano-composite screening
- healthy witnesses: fourteen healthy witnesses who have never been in contact with lightning, matched on age and sex
  Interventions: Diagnostic Test: nano-composite screening

INTERVENTIONS:
Diagnostic Test: nano-composite screening — Recovery of the bottoms of the victims' blood and urine tubes at H+4. Blood and urine samples from the victims at two years of age. Single blood and urine samples from the witnesses

SUMMARY:
Objective: To demonstrate the presence of bioresistant intracorporeal carbon-based nanocomposites in subjects exposed to a fulguration, in the immediate aftermath of this fulguration and 24 months (+/- 6 months) after the accident, on blood and urine samples, then in comparison with blood and urine samples from 14 healthy subjects.

Hypothesis: Lightning discharge in the human body reveals the presence of multi-functional nanoparticles which are reassembled under the impact of the electric discharge into nanostructured films, filaments and aggregates; they consist of dispersed graphene-like nanoparticles embedded in an aliphatic cross-reticulated matrix. The high electrical conductivity of the nanoinclusions, their refractory properties and the cross-reticulation of the nanoassemblages explain their biorésistance.

The graphene-like multi-functional nanoparticles are assumed to trace a population of aerosols formed in the atmosphere by plasma discharge which is present in air, water and all natural resources. Their ability to undergo changes from folded nanosheets to confined ultra-fine nanoparticles allow them to be inhaled or absorbed by the human body, or to be ingested with food.

DETAILED DESCRIPTION:
In order to detect nanocomposites in patients who have been impacted by lightning, an analysis protocol will be performed on the remains of blood and urine samples from their initial medical admission. After filtering the blood and urine samples, the remaining nanocomposites are selected for characterization, at micro to nanoscale, using the scanning electron microscope and the transmission electron microscope.

Based on laboratory experiments, a second sampling of blood and urine will be performed 24 months (+/-6 months) after the lightning strike to follow the delayed production of nanocomposites from the remaining activated nanoparticles.

* Presence of bioresistant nanocomposites in blood and urine at D0 and M24 (+/- 6 months) :
* If the victim was treated between H0 and H2 after the fulguration : an initial blood sample was taken by the SMUR or the emergency room and stored
* If the victim was treated between H0 and H6: urine sample was taken from the first urine after fulguration.
* At M24 (+/- 6 months) after the fulguration: collection of 18 ml of blood and two bottles of urine.

In order to describe the neurological disorders of the patients, initial clinical, biological and radiological data will be collected in the patients' medical records and a new clinical examination will be performed at 24 months (+/- 6 months) after fulguration.

-Search for descriptive data.

1. testimonials

   Data collected:

   - During the interrogation of the patient on the day of the fulguration
   * In the medical file of the patient consulted at the department's administration
   * During the interview organized at 24 months (+/- 6 months) after the fulguration
   * Entry in the observation logbook (RedCap)
2. clinics

   Data collected :
   * From the day of the fulguration, in the medical file of the patient consulted at the department's administration
   * During the interview organized at 24 months (+/- 6 months) from the fulguration where a clinical examination will be carried out.
   * Entry in the observation notebook (RedCap)
3. organic

   Data collected :
   * In the medical record of the patient at the time of the fulguration consulted at the department's administration
   * from biological samples taken 24 months (+/- 6 months) after fulguration
   * Entry in the observation logbook (RedCap)
4. imagery

   Data collected :

   - In the medical file of the patient consulted at the department's administration
   * Entry in the observation logbook (RedCap)
   * Presence and description of neurological disorders in exposed patients, immediately after the event and M24 (+/- 6 months) after the accident.

   H0 will be the time when the accident took place. H0-H12: Collection of clinical, biological and radiological information in the patient's medical record. Recovery at M24 (+/- 6 months) for immediate or prolonged initial neurological disorders.

   At M24 (+/- 6 months): medical examination at the patient's home to :
   * hear their testimony
   * describe the delayed neurological disorders This interview will be based on the Toulouse fulgurate questionnaire.
   * Description of the treatments administered to the exposed patients during the 2 years following the accident (medication, physiotherapy, rehabilitation, work stoppage).
   * Depending on their complaints, patients will be taken care of by various health professionals (general practitioner, physician, pharmacist, physiotherapist, occupational therapist, speech therapist) who will prescribe various types of care (medication, leave from work, physiotherapy, rehabilitation).
   * At M24 (+/- 6 months), after questioning the patient and his doctor, the care received will be traced (qualitative and quantitative).
   * Descriptions of the effects of the treatments administered during the 2 years following the accident.

   At M24 (+/- 6 months): Description of the evolution of neurological disorders in time, recovery quality and location.

   - Presence and description of other organic lesions.

   - The objective is to know what other internal organs may have been affected by the lightning strike

   - Looking through the medical file for the clinical examination of J0 and those of follow-ups
   * Looking through the biological assessment carried out immediately after the event between H0 and H12 in the lighting-stroke patient to highlight which organs were affected (bloodlines, kidney, liver, muscle, heart).
   * Basic biology screening to look for the following information:
   * NFS / Platelet / VS / Coagulation check-up
   * Blood ionogram (Na+ Cl- K+ Total Ca ionized Ca Mg++ HCO3- HPO4--)
   * Blood creatinine / urea / CPK / LDH
   * Troponin in cycle
   * Liver check-up
   * CRP

   Description of measures taken to reduce and avoid bias

   Measurement bias:
   * Preliminary experiments carried out by the CNRS team with a lightning reactor on self-samples of urine in order to obtain comparative images, adapt the manipulations and anticipate the preparation of the lighting-stroke patient samples to select the most representative nanocomposites for high resolution microscopic characterization.
   * During the analysis of the samples, the only two experimenters will be the investigator coordinating the study, Dr FOUSSAT, and Dr COURTY. There will be a double reading of each sample with consultation on the description.
   * Photos will be taken with the same camera.

   Selection bias:

   - None, because all 14 patients were fulgurated.

   Memory bias:

   - Cross-check the patients' testimonies with the analyses and complementary examinations carried out, requested by the attending physician or another health professional.

   Sampling bias:

   - Matching the 14 healthy subjects to the age and sex of the 14 fulgurated subjects.

   In order to better understand the mechanisms of in vivo formation of these nanocomposites, an attempt will be made to identify them in healthy subjects.

   -Qualitative and quantitative aspects of bioremediation nanocomposites possibly identified in the blood of subjects not affected by lightning-strike.

   Analysis of the blood of 14 healthy patients for:
   * controlling stochastic forming mechanisms of polymer nanocomposite;
   * controlling effects of environmental factors (air and water quality) on the abundance and properties of airmade polymer nanocomposites
   * proof-of-concept justification
   * full analytical procedure.

   Low levels of bioresistant nanocomposites are expected in this group. The aim is to trace the occurrence of nanocomposites formed by plasma discharges in the atmosphere which have passed through the alveolar and digestive barrier into the bloodstream.

   The blood of healthy subjects will be collected at the Aurillac CH laboratory by taking an additional 18 ml on sodium heparinate tube during a blood test for routine check-up (INR monitoring for example). Patients will be given an information note and a consent form stating that they accept this additional volume of sample. They will inform their work and their commune of residence.

   The samples will be anonymised and packaged for transport to the Aurillac laboratory for analysis under a stereomicroscope microscope in the alcoholic liquid phase. They will then be sent in dry form to the CNRS for analysis by scanning and transmission electron microscope.

ELIGIBILITY:
Inclusion criteria :

-Patients exposed: all subjects who were victims of the fulguration accident.

Non-exposed patients:

* 14 subjects,
* of all ages,
* free of major pathology and having never been the victim of a fulguration accident, nor having witnessed a fulguration at less than 20 meters,
* having never worked in a high-energy environment (CEA, EDF, particle accelerator, AREVA-type laboratory, radiology manipulator, radiation protection profession).

Exclusion criteria :

* Pregnant or breastfeeding woman.
* Subject under guardianship, curatorship or safeguard of justice, or deprived of liberties.
* Any condition judged by the investigator to be incompatible with the research.
* Refusal to participate. Exposed patients: if the above-mentioned accident induced more than a simple lightning strike (lightning: died by lightning, electrocution: touched by an electric current, electrocution: died by contact with an electric current).

Ages: 7 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients affected by lightning in collective fulguration and healthy witnesses who have never been in contact with lightning, matched on age and sex
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Description of bioresistant nanocomposites | Day 0
  Characterization in blood
Description of bioresistant nanocomposites | Month 24
  Characterization in blood
Description of bioresistant nanocomposites | Hour 12
  Characterization in urine
Description of bioresistant nanocomposites | Month 24
  Characterization in urine

SECONDARY OUTCOMES:
neurological disorders | Day 0
  Research and description of neurological disorders with questioning of date of onset and duration
neurological disorders | Month 24
  Research and description of neurological disorders with questioning of date of onset and duration
neuropsychological disorders | Day 0
  Research and description of neuropsychological disorders with questioning of date of onset and duration
neuropsychological disorders | Month 24
  Research and description of neuropsychological disorders with questioning of date of onset and duration

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Caumon, Principal Investigator — CH Henri Mondor (Aurillac)
Locations (5):
- France (5):
  - CH Henri Mondor, Aurillac
  - CH de Luneville, Lunéville
  - CHRU Bradois, Nancy
  - CHRU de Nancy, Nancy
  - CH de SAINT-DIE-DES-VOSGES, Saint-Dié

IPD SHARING:
Plan to Share IPD: Undecided